CLINICAL TRIAL: NCT01890577
Title: An Observational Study of South African Dialysis Patients Treated With Aranesp
Brief Title: Study of South African Dialysis Patients
Status: Terminated | Type: Observational
Why Stopped: Study was terminated due to slow enrolment with no reasonable expectation of attaining a meaningful sample size
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20110243
Record Dates: First submitted 2013-04-18; First posted 2013-07-02 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Chronic Kidney Disease, Receiving Dialysis
Keywords: Chronic kidney disease; Dialysis; Erythropoiesis stimulating agent; South Africa
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Darbepoetin alfa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study population: Single cohort of dialysis patients
  Interventions: Drug: Aranesp

INTERVENTIONS:
Drug: Aranesp — Observational study; minimum single dose of Aranesp required for eligibility; no protocol-specified regimen; study must not influence normal clinical practice.

SUMMARY:
An observational study to describe the treatment of anaemia in patients with chronic kidney disease, who are receiving dialysis treatment at selected study centres in South Africa.

DETAILED DESCRIPTION:
This multicentre, prospective, observational study will describe the treatment and clinical outcomes of of dialysis patients in South Africa. No formal hypothesis will be tested in this descriptive study. Eligible subjects will be receiving either peritoneal or haemodialysis, will have received Aranesp therapy between 3 and 6 months prior to enrolment into the study, do not need to be receiving Aranesp at the time of enrolment and will be followed for up to 12 months after commencement of Aranesp. Data to be collected includes ESA therapies, iron usage, relevant concomitant therapies, haemoglobin concentrations, other relevant clinical laboratory parameters and red cell transfusions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing chronic haemodialysis or peritoneal dialysis
* Commenced Aranesp therapy 3-6 months prior to enrolment
* Erythropoiesis stimulating agent (ESA) naive or treated with another ESA prior to commencing Aranesp
* Informed consent obtained

Exclusion Criteria:

* Received Aranesp in an interventional study within 6 months prior to start of observation period
* Receive investigational product during the observation period

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients receiving dialyis at South African study centres and having received at least one dose of Aranesp
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (7):
- South Africa (7):
  - Research Site, Glenwood, KwaZulu-Natal
  - Research Site, Umhlanga, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
  - Research Site, Durban
  - Research Site, Kimberley
  - Research Site, Lenasia
  - Research Site, Roodepoort

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Aranesp®: Participants receiving Aranesp® (darbepoetin alfa) for at least 3 months prior to enrolment and according to the local prescribing guidelines.
Period: Overall Study
Arm/Group | Aranesp®
Started | 28
Completed | 0
Not Completed | 28

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) consists of all patients enrolled into the study after commencing Aranesp® therapy amd with reported data
Arm/Group | Aranesp®
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] — Age data were available for 27 participants
  years | 55.8 (15.1)
Gender [Number; unit: participants] — Gender data were available for 27 participants
  participants
    Female | 13
    Male | 14
Race/Ethnicity, Customized [Number; unit: participants] — Race data were available for 27 participants
  participants
    White/caucasian | 1
    Black | 12
    Asian | 11
    Colored | 3
Baseline Hemoglobin Concentration [Mean (Standard Deviation); unit: g/dL] — Data were available for 11 participants
  g/dL | 9.7 (2.0)
Baseline Aranesp Route [Number; unit: participants]
  Intravenous | 1
  Subcutaneous | 27
Baseline Aranesp Dose [Mean (Standard Deviation); unit: µg/week] | 36.6 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Haemoglobin Concentration
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Each 4-week period for the duration of the study period (15 months)
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

2. Secondary Outcome: Hemoglobin Excursions
Description: Hemoglobin excursions defined as hemoglobin <10g/dL and >12g/dL. Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

3. Secondary Outcome: Hemoglobin Within the Range 10-12 g/dL Over Time
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: On a continuous basis over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

4. Secondary Outcome: Erythropoiesis Stimulating Agent (ESA) Usage
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

5. Secondary Outcome: ESA/Aranesp Dose Ratio
Description: Ratio of the calculated mean weekly dose equivalent of an ESA administered immediately prior to conversion to treatment with Aranesp, to the calculated mean weekly dose equivalent of the first dose of Aranesp administered at commencement. Not applicable to participants who were ESA-naive at time of Aranesp commencement.
  Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Day of commencement of Aranesp
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

6. Secondary Outcome: Iron Therapy Use
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

7. Secondary Outcome: Use of Concomitant Therapies: Immunosuppressants, Cardiovascular Medications, Secondary Hypoparathyroidism Medications, Anti-retroviral Therapy
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: At each 12-week interval over the observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

8. Secondary Outcome: C-Reactive Protein, Albumin, Transferrin Saturation and Serum Ferritin Concentration
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Red Blood Cell Transfusions
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Hospitalisations
Description: Due to the premature termination of the study no outcome measure data were analyzed.
Time Frame: Over the 15-month observation period
Arm/Group | Aranesp®
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 15 months
Description: Only serious and non-serious adverse drug reactions which in the Investigator's opinion are causally related to Aranesp were collected during this observational study.
Arm/Group | Aranesp®
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.